CLINICAL TRIAL: NCT00427856
Title: A Multi-Center, Open-Label, Phase II Study of Sequential, Single-Agent Obatoclax Mesylate (GX15-070MS)Followed by a Combination With Rituximab to Patients With Previously-Untreated Follicular Lymphoma (FL)
Brief Title: Safety and Efficacy of Single Agent Obatoclax Mesylate (GX15-070MS) Followed by a Combination With Rituximab for Previously-untreated Follicular Lymphoma (FL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM014
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obatoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obatoclax mesylate 40mg (Experimental): 40 mg over 3 hrs q/weekly for 12 weeks, 4 weeks combo with rituximab, another 8 weeks single-agent obatoclax
  Interventions: Drug: Obatoclax mesylate; Drug: Rituximab
- Obatoclax mesylate 60mg (Experimental): 60 mg obatoclax mesylate over 24 hours, q/weekly for 12 weeks, 4 weeks combo with rituximab, another 8 weeks single-agent obatoclax
  Interventions: Drug: Obatoclax mesylate; Drug: Rituximab

INTERVENTIONS:
Drug: Obatoclax mesylate — Obatoclax mesylate 40mg, and 60mg
  Other Names: (GX15-070MS)
Drug: Rituximab — Rituximab

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogenic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase II study of obatoclax administered alone as a weekly, 3-hour or 24-hour infusion for 12 weeks followed by a combination with rituximab to patients with previously-untreated Follicular Lymphoma. For purposes of clinical evaluations, treatment cycles will occur in 4-week periods. Treatment may be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described may be administered with the intent to treat the patient's malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of Follicular Lymphoma (FL)
* Must have advanced stage disease
* Must not have received any prior chemotherapy or immunotherapy for lymphoma, including steroids
* Must have adequate organ function
* Must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Response rate | 12 weeks

SECONDARY OUTCOMES:
Time to Tumor Progression. | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (1):
- The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States